CLINICAL TRIAL: NCT04457193
Title: Outcomes After Transoral Incisionless Fundoplication (TIF) Following Successful Endoscopic Ablation for Barrett's Esophagus: A Pilot Study
Brief Title: Outcomes After Transoral Incisionless Fundoplication (TIF) Following Successful Endoscopic Ablation for Barrett's Esophagus
Status: Enrolling by invitation | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00164823
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Barrett Esophagus; Transoral Incisionless Fundoplication
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- post-ablation Barrett's patients: The patients with known prior diagnosis of histologically-confirmed Barrett's esophagus with or without dysplasia who have documentation of complete remission of Barrett's esophagus by endoscopy and histology after endoscopic ablation
  Interventions: Device: TIF

INTERVENTIONS:
Device: TIF — Transoral Incisionless Fundoplication (TIF) is an endoscopic procedure that mechanically creates fundoplication similar to traditional operative Nissen fundoplication. The role of TIF in patients with BE whom underwent successful endoscopic ablation has not been fully investigated.

SUMMARY:
Barrett's esophagus (BE) is a precancerous lesion characterized by the replacement of the normal stratified squamous epithelium of the distal esophagus by intestinal metaplasia (IM). Non-dysplastic BE may progress to low-grade dysplasia (LGD), to high-grade dysplasia (HGD) and esophageal adenocarcinoma (EAC). Endoscopic ablation is safe and effective for complete eradication of BE. However, recurrence is common. Cumulative incidence rate of BE recurrence is up to 30% in the third year. Thus, achieving complete eradication of IM, patients should undergo surveillance indefinitely with serial endoscopy to assess for recurrence of BE. In addition, BE patients have been committed to life-long proton pump inhibitor (PPI) therapy, but increasing concerns about adverse effects has led to alternative therapies. Studies have showed that laparoscopic Nissen fundoplication may decrease recurrence of BE after endoscopic ablation. Transoral Incisionless Fundoplication (TIF) is an endoscopic procedure that mechanically creates fundoplication similar to traditional operative Nissen fundoplication. The role of TIF in patients with BE whom underwent successful endoscopic ablation has not been fully investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years
* Known prior diagnosis of histologically-confirmed BE with or without dysplasia (as defined by the presence of specialized columnar epithelium anywhere in the tubular esophagus with >= 1 cm of circumferential involvement or non-circumferential involvement of specialized columnar epithelium) [Prague class >1] and history of initial complete eradication-IM following endoscopic ablation for Barrett's esophagus.
* Documentation of complete ablation of BE by endoscopy and histology after radiofrequency or cryotherapy ablation on two endoscopic examinations at least 3 months apart, within most recent endoscopy performed within 6 months. Pathologic diagnosis determined by the expert pathologist at each site.
* On PPI therapy, who opt for an intervention over lifelong drug dependence.
* Hiatal hernia ≤ 2 cm or Hill grade < 2 [unless patients undergoing combined TIF and hiatal hernia repair]
* Abnormal esophageal acid exposure [Percent esophageal acid exposure time > 6% defined by Bravo ph monitoring (48 - 96 hours study)
* Able to provide informed consent

Exclusion Criteria:

* Age < 18 or > 75 years
* Inability to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with history Barrett's esophagus who have resolution of Barrett's mucosa after endoscopic ablation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-06-07 (Actual); Primary Completion 2027-06-07 (Estimated); Study Completion 2027-06-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with normal esophageal acid exposure time | 6 months
  Normal esophageal acid exposure time is 6 percent or less.

SECONDARY OUTCOMES:
Percentage of participants that are able to discontinue PPI post TIF | 6 months
  Percentage of participants that are able to discontinue PPI post TIF will be assessed at 6 months.
Incidence of esophagitis post-TIF | 6 months
  The presence of esophagitis on upper endoscopy.
Proportion of patients with recurrence of BE and BE-related dysplasia | Up to 36 months
  Proportion of patients with recurrence of BE and BE-related dysplasia will be assessed up to 36 months.
Number of TIF-related serious adverse events | Up to 36 months
  Treatment related serious adverse events (SAEs) including hospitalization, unscheduled emergency room or physician visits for post-TIF symptoms), bloating, dysphagia.
Change in quality of life as assessed by the GERD-Health-related quality of life Questionnaire | Baseline, 6, 12, 24 and 36 months
  The GERD-Health-related quality of life (HRQL) Questionnaire has an overall score range of 0 to 75. Each item is scored from 0 to 5, with a higher score indicating worse symptoms and poorer quality of life.
Change in Gastroesophageal Reflux Disease (GERD) symptoms assessed by the Reflux Symptom Index (RSI) | Baseline, 6, 12, 24 and 36 months
  The RSI is a nine-item self-administered outcome questionnaire designed to document reflux symptoms and severity. Each item is scored on a scale of 0 (no problem) to 5 (severe problem), with overall score ranging between 0 and 45. Higher scores mean more severe symptoms. RSI > 13 may be indicative of significant reflux disease.

CONTACTS AND LOCATIONS:
Overall Officials: Saowanee Ngamruengphong, Principal Investigator — Johns Hopkins University
Locations (1):
- Saowanee Ngamruengphong, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No